CLINICAL TRIAL: NCT02294669
Title: A Feasibility Study to Evaluate the TURRIS Facet Fusion System as an Adjuvant to Unilateral Pedicle Screw Fixation in Lumbar Spinal Surgery
Brief Title: A Feasibility Study to Evaluate the TURRIS Facet Fusion System in Lumbar Spinal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Strategic reasons
Sponsor: SpineWelding AG (Industry)
Collaborators: ISS integrated Scientific Services AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Turris
Record Dates: First submitted 2014-11-03; First posted 2014-11-19 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Spinal Disease
MeSH Terms: conditions — Spinal Diseases

ARMS (1):
- Turris Facet Fuser (Experimental)
  Interventions: Device: Turris Facet Fuser

INTERVENTIONS:
Device: Turris Facet Fuser — Study participants will have a Turris Facet Fuser inserted into the contralateral facet joint, instead of a state of the art contralateral pedicle screw system.

SUMMARY:
This is a prospective, exploratory study to verify intra-operative handling and safety and to collect preliminary short-term safety and efficacy data of the Turris® Facet Fuser, a small bioresorbable device for the immediate immobilization of the facet joint.

Patients eligible for study enrollment will present with degenerative lumbar spinal diseases involving the L4/L5 segment and requiring spinal fusion.

DETAILED DESCRIPTION:
The Turris® Facet Fuser is an investigational resorbable device intended to support spinal segment fusion in individuals suffering from degenerative lumbar spinal diseases. The device is directly inserted in the facet joint of the affected segment using the BoneWelding® technology, a soft tissue sparing, ultrasound based insertion method which confers immediate stability to the implant.

Aim of this prospective, exploratory study is to verify intra-operative handling and safety of the Turris® Facet Fusion System and to collect preliminary short-term safety and efficacy data on this innovative implant by observing the healing process over a period of one year.

ELIGIBILITY:
Inclusion Criteria:

* one-level fusion at L4/L5 with dorsal instrumentation and, if required, with monolateral decompression and/or intervertebral disc removal and implantation of an intervertebral implant

Exclusion Criteria:

Patient

* had previous surgical stabilizations at the involved or adjacent levels
* has lytic spondylolisthesis
* has degenerative spondylolisthesis grade II or higher
* has radiographic signs of significant instability and/or hypermobility of the segment (>3mm translation, >11° rotation difference from adjacent level)
* has scoliosis > 10° at the involved segment
* has osteoporosis to a degree that spinal instrumentation would be contraindicated.
* has presence of active malignancy.
* has overt or active infection, either local or systemic
* is less than 18 years old
* is pregnant or plan a pregnancy during the study duration
* has a BMI > 35
* has a progressive neuromuscular disease
* has a condition which requires postoperative medications that may interfere with bone metabolism
* has a history of autoimmune disease
* has a history of endocrine or metabolic disorders known to affect osteogenesis
* is mentally ill or incompetent
* is an alcohol and/or drug abuser
* is not available for follow up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-06-18 (Actual); Study Completion 2016-06-18 (Actual)

PRIMARY OUTCOMES:
The number, severity and causality of intra-operative and post-operative complications | 1 year
  Patients will be observed during hospitalization, at 6 weeks, 3 months, 6 months and 12 months

SECONDARY OUTCOMES:
Fusion of the L4/L5 Segment | within 12 months
Change from Baseline in Spine Tango Oswestry score | Baseline, 3 months, 6 months and 12 months
Change from Baseline in Spine Tango COMI score | Baseline, 3 months, 6 months and 12 months
Change from Baseline in Spine Tango VAS score for back- and leg-pain | Baseline, 3 months, 6 months and 12 months
Intraoperative radiation exposure | intra-operative
  Radiation exposure time during the insertion process of the pedicle screw system and the Turris Facet Fusion will be recorded separately

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Berlemann, MD, Principal Investigator — Rückenzentrum Oberaargau
Locations (2):
- Switzerland (2):
  - Neuro- und Wirbelsäulenzentrum, Cham, CH
  - Rückenzentrum Oberaargau AG, Langenthal